CLINICAL TRIAL: NCT07339709
Title: Intraperitoneal Pressure Measurements Survey in Pediatric Centers
Acronym: IPP
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9764
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Renal Failure
Keywords: Pediatric Renal Failure; Peritoneal dialysis; Intraperitoneal pressure; Intraperitoneal dialysates; End-stage renal disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intraperitoneal pressure (IPP) is an objective measurement used to assess tolerance to fluid volume. IPP has been shown to be strongly correlated with intraperitoneal dialysate volume as well as anthropometric parameters. In observational studies conducted in adults, an IPP greater than 13-14 cmH2O was associated with an increased risk of peritonitis, initiation of hemodialysis, or death.

Measuring IPP is therefore a tool to optimize dialysis prescriptions. However, this measurement is not well standardized, and there is limited scientific evidence regarding its impact on patient management.

Measuring IPP is a tool to optimize dialysis prescriptions. However, this measurement is not well standardized, and there is limited scientific evidence regarding its impact on patient management. Some centers do not perform any measurements, others perform them monthly, and some only during peritoneal equilibration tests.

The hypothesis of this research is to highlight current practices and experiences in measuring intraperitoneal pressures in children undergoing peritoneal dialysis in different European dialysis centers, in order to improve practices regarding PIP prescription.

ELIGIBILITY:
Inclusion Criteria:

- Healthcare professional working in a European dialysis center

Exclusion Criteria:

- Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthcare professional working in a European dialysis center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07-16 (Estimated)

PRIMARY OUTCOMES:
Review of current practices in measuring intraperitoneal pressures in children undergoing peritoneal dialysis | Up to 12 months
  This study aims to provide an overview of current experiences in measuring intraperitoneal pressures in children undergoing peritoneal dialysis in different European dialysis centers.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de pédiatrie 1 - CHU de Strasbourg - France, Strasbourg, France